CLINICAL TRIAL: NCT04135976
Title: Applicability of the International Classification of Functioning, Disability and Health (ICF) in Primary Care Physiotherapy Units in the Health Service of Castille and Leon (Spain)
Brief Title: Applicability of the ICF in Primary Care Physiotherapy Units in the Health Service of Castille and Leon (Spain)
Status: Completed | Type: Observational
Sponsor: University of Valladolid (Other)
Collaborators: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Héctor Hernández Lázaro, Principal investigator, University of Valladolid
Other Study IDs: CEIC 2231
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: physiotherapy; primary health care; ICF; core set validation; musculoskeletal conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary care physiotherapy units of the Spanish health service in Castille and Leon (SACYL) are responsible for providing physiotherapy treatments to the general population. Being part of the primary health care system, the actions of these units are aimed at the treatment of common conditions that do not involve severity, frequently musculoskeletal disorders.

The work of physiotherapists is closely related to the functionality of patients and, in this sense, the World Health Organization (WHO) has proposed the International Classification of Functioning, Disability and Health (ICF) as a conceptual framework to characterize the functional status of individuals.

The use of ICF in the clinical setting is not sufficiently widespread due to the the difficulties that the use of such an exhaustive classification implies in practice. In an attempt to address this problem, the WHO has encouraged the development of reduced versions aimed at responding to specific conditions or care contexts.

The idea behind the development of core sets is that it is possible to select a number of categories so as to capture the essence of a given clinical process, allowing an agile use of the ICF. However, in order to put these core sets into practice, it is necessary to check that the selected categories are valid from the perspective of the participants in the clinical processes.

The purpose of this research project is to determine whether the musculoskeletal core sets of the ICF are applicable in SACYL primary care physiotherapy units. This implies knowing if the categories already selected in these sets are representative of the health aspects considered as most relevant in the clinical context of physiotherapy in primary care.

To achieve this, four studies will be conducted to capture the perspective of patients, physiotherapists, researchers and clinical practice. This information will be translated into the language of the ICF to obtain comparable categories with those present in the core sets.

In this way, this research project will make possible to validate or adapt the core sets of the ICF for musculoskeletal conditions, in a specific clinical context of physiotherapy in primary care.

DETAILED DESCRIPTION:
Preliminary studies will attempt to capture the perspectives of all agents involved in the SACYL primary care physiotherapy clinical processes.

The perspective of the patients will be collected by means of a qualitative study through focal groups of people who have been attended in physiotherapy units in primary care. Each focus group will be made up of five patients who will be provided with information about the ICF and will be encouraged to express themselves on the aspects that they consider most relevant when they are attended in primary care physiotherapy units. The duration of these focus groups will be 30 minutes and as many groups as necessary will be conducted to reach 100% saturation. The information obtained will be translated into second level categories of the ICF, so that it can be compared with those present in the already existing core sets.

The perspective of the physiotherapists will be gathered through a Delphi study. Physiotherapists with experience in the care context under study will be selected and the information will be collected through online surveys. Three rounds will be carried out, translating the information obtained into second level categories of the ICF, and providing feedback in each round to the participants.

The research perspective will be studied through a systematic review of the scientific literature. To this end, the main databases will be scrutinized and studies that investigate musculoskeletal conditions will be selected in a context compatible with that of physiotherapy in primary care. The data will be obtained through the outcome measures used in these studies, including those with an agreement level equal to or greater than 5%. This information will be translated into second level categories of the ICF, allowing us to know which of them are more relevant.

The clinical point of view will be captured in a transversal study in which a sample of patients receiving physiotherapy services in primary care will be taken. These patients must make an assessment of the categories present in the ICF checklist. This list will be complemented with the categories of the core sets for musculoskeletal conditions and with those detected in the previous studies. The participants will assign a qualifier to each category, depending on the importance they attach to it. In this study, patients will also be assessed using a generic test that measures the degree of functionality. Aspects such as the presence of cognitive deficit, depression and quality of life will also be considered. The measurement instruments will be selected from the results obtained in the bibliographic review described above. The number of patients required is estimated at 50 individuals belonging to different basic health areas. The data obtained will be analysed and translated into the language of the ICF (second level categories).

The categories derived from the set of previous studies will be compared with those present in the core sets of the ICF for musculoskeletal conditions. Three types of results are expected to be obtained: categories coincident in both groups of data, categories detected in the studies carried out but absent in the core sets; and categories not detected but present in the core sets.

In this way, it will be possible to determine the best way to establish the use of the ICF in the primary care physiotherapy units of SACYL.

ELIGIBILITY:
Systematic review:

* Inclusion Criteria:
* Primary care studies over adult general population in developed Western countries
* Published in a peer-review journal
* Published since 2009
* Type of publication: random controlled trials, controlled clinical trial, cross-sectional study, observational study and qualitative study
* Exclusion Criteria:
* Studies based solely in specific health problems
* Studies not conducted over general population (some kind of selection based on ethnicity, sex, social class, etc. have been made).
* Studies with hospitalized participants
* Studies published in a language other than English or Spanish

Expert survey:

* Inclusion Criteria:
* Physiotherapists with at least two years of professional experience in primary health care.

Qualitative study

* Inclusion Criteria:
* Treated in a physiotherapy unit during the past year.
* Over 18 years old
* Exclusion Criteria:
* Inability to concentrate for 30 minutes.
* Insufficient knowledge of the Spanish language.

Empirical multicenter study:

* Inclusion Criteria:
* Patients over 18 years referred to a primary care physiotherapy unit
* Exclusion Criteria:
* Inability to concentrate for 30 minutes.
* Insufficient knowledge of the Spanish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population over 18 years of age that has been treated in a physiotherapy unit in primary care during the last year, or is going to be treated in these units during the development of this research project.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Most important issues related to functional status, disability and health in the treatment of musculoskeletal conditions in primary care, according to the ICF, reported in the scientific literature. | 2022/05 - 2022/09
  The measurement instruments used by primary care researchers will be broken down into units of meaning and converted into ICF categories using the conversion rules proposed by Cieza et al. The primary result is the achievement of the categories considered most relevant by primary care researchers.
Most important issues related to functional status, disability and health in general population treated in physical therapy units for musculoskeletal conditions reported by physiotherapists in an online survey (expert survey). | 2020/06 - 2021/03
  The primary outcome will be a set of ICF categories that will be representative of the physiotherapists' perspective. The Delphy study will gather information from physioterapists working in a primary care set. This information will be converted into ICF categories using the conversion rules.
Most important issues related to functional status, disability and health in general population treated in physical therapy units for musculoskeletal conditions reported by these patients in focus groups (qualitative study). | 2022/05 - 2022/12
  The primary outcome will be a set of ICF categories that will be representative of the patients' perspective. The focus groups will provide information about the point of view of the patients treated in primary care physioterapy units. Using the conversion rules, the information will be translated into ICF categories.
Most important issues related to functional status, disability and health in patients treated in physical therapy units for musculoskeletal conditions, assessed by the comprehensive musculoskeletal ICF core set (empirical multicenter study). | 2022/05 - 2023/03
  Physiotherapists will evaluate a group of patients using the comprehensive ICF core set for post-acute musculoskeletal conditions. These patients will be asked to assess the relevance of the categories included in the ICF core set, according to their health problem. A 0-100 mm visual analog scale (VAS) will be used to rate each ICF category (a score of 5 or higher would validate the ICF category). The primary outcome will be the percentage of validated categories included in the ICF core set.

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Mingo Gómez, Study Director — University of Valladolid; Héctor Hernández Lázaro, Principal Investigator — University of Valladolid; Sandra Jiménez del Barrio, Study Director — University of Valladolid; Luis Ceballos Laita, Study Director — University of Valladolid
Locations (1):
- Ólvega Primary Health Center, Ólvega, Soria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hernandez-Lazaro H, Mingo-Gomez MT, Ceballos-Laita L, Medrano-de-la-Fuente R, Jimenez-Del Barrio S. Validation of the international classification of functioning, disability, and health (ICF) core sets for musculoskeletal conditions in a primary health care setting from physiotherapists' perspective using the Delphi method. Disabil Rehabil. 2023 Jul;45(15):2458-2468. doi: 10.1080/09638288.2022.2096128. Epub 2022 Jul 13. PMID 35830343
- [Result] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Lahuerta-Martin S, Hernando-Garijo I, Medrano-de-la-Fuente R, Ceballos-Laita L. Researcher's Perspective on Musculoskeletal Conditions in Primary Care Physiotherapy Units through the International Classification of Functioning, Disability, and Health (ICF): A Scoping Review. Biomedicines. 2023 Jan 20;11(2):290. doi: 10.3390/biomedicines11020290. PMID 36830831
- [Result] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Rodriguez-Fernandez AI, Areso-Boveda PB, Ceballos-Laita L. Validation of the International Classification of Functioning, Disability, and Health (ICF) core set for post-acute musculoskeletal conditions in a primary care physiotherapy setting from the perspective of patients using focus groups. Disabil Rehabil. 2024 Aug;46(16):3594-3601. doi: 10.1080/09638288.2023.2251392. Epub 2023 Sep 5. PMID 37667886
- [Result] Hernandez-Lazaro H, Jimenez-Del Barrio S, Ceballos-Laita L, Lahuerta-Martin S, Medrano-de-la-Fuente R, Hernando-Garijo I, Mingo-Gomez MT. Multicentre cross-sectional study assessing content validity of the International Classification of Functioning, disability and health core set for post-acute musculoskeletal conditions in primary care physiotherapy services. J Rehabil Med. 2023 Nov 16;55:jrm11950. doi: 10.2340/jrm.v55.11950. PMID 37974517